CLINICAL TRIAL: NCT04036435
Title: An Open-Label, Multi-Center Extension Study to Characterize the Long-Term Safety and Efficacy of BMS-986165 in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: Long-Term Study That Measures the Safety and Efficacy of Deucravacitinib (BMS-986165) in Participants With Psoriasis
Acronym: POETYK PSO-LTE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-075; 2019-000612-29 (Registry Identifier: EudraCT)
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986165 (Experimental)
  Interventions: Drug: BMS-986165
- Vaccine Cohort (Experimental)
  Interventions: Drug: BMS-986165; Drug: Placebo

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Other Names: Deucravacitinib
Drug: Placebo — Specified dose on specified days
  Arms: Vaccine Cohort

SUMMARY:
The main purpose of this study is to evaluate the long-term safety and efficacy of the drug Deucravacitinib (BMS-986165) in participants who have been previously enrolled in an applicable Phase 3 psoriasis study. In addition, the study includes a vaccine cohort to evaluate whether deucravacitinib impacts the humoral immune response to 2 non-live vaccines, the Pneumovax 23 vaccine (pneumococcus), a T-cell independent vaccine, and the Boostrix vaccine (tetanus toxoid), a T-cell dependent vaccine. Additionally, this vaccine cohort assesses the safety of administering these vaccines to subjects with psoriasis receiving deucravacitinib compared to those receiving a placebo.

ELIGIBILITY:
Inclusion Criteria

* Completion of the protocol-required treatment period in an applicable study of BMS-986165 in moderate-to-severe psoriasis.
* Women must not be pregnant, lactating, or breastfeeding.
* Vaccine Cohort:

  1. Subject must have moderate-to-severe plaque psoriasis, be currently receiving deucravacitinib treatment in the main IM011075 LTE cohort in the United States, Canada, or Poland, and must have completed at least one year of deucravacitinib treatment.

Exclusion Criteria

* Any disease or medical condition that the investigator feels that would make the patient unsuitable for this study.
* To be eligible for the study, a participant must not have active signs or symptoms of tuberculosis (TB) as judged by the investigator.
* Vaccine Cohort:

  1. Subject received the Pneumovax 23 vaccine ≤ 5 years before Day 1 or a pneumococcal conjugate vaccine ≤ 1 year before Day 1.
  2. Subject received the Boostrix vaccine (as single or part of a combination vaccine) ≤ 5 years before Day 1.
* Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1466 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-07-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 244 weeks
Incidence of Serious Adverse Events (SAEs) | Up to 244 weeks
Proportion of participants achieving a satisfactory humoral response: pneumococcus | At Week 4 post vaccination
  Vaccine cohort only
  Defined as ≥ 2-fold increase in immunoglobulin (IgG) antibody titers or geometric mean fold rise (GMFRs) titers of ≥ 6
Proportion of participants achieving a satisfactory humoral response: tetanus titers | At Week 4 post vaccination
  Vaccine cohort only
  A serologic response is defined as:
  * Postvaccination titer levels ≥ 0.40 IU/mL if prevaccination IgG antibody titer level is ≤ 0.10 IU/mL OR
  * Postvaccination titer levels of at least a 4-fold increase if prevaccination titer level is > 0.10 IU/mL and ≤ 2.7 IU/mL OR
  * Postvaccination titer levels of at least a 2-fold increase if prevaccination titer level is > 2.7 IU/mL

SECONDARY OUTCOMES:
static Physician Global Assessment (sPGA) 0/1 response | Up to 240 weeks
Psoriasis Area and Severity Index (PASI) 75 response | Up to 240 weeks
Proportion of participants with anti-tetanus toxoid IgG geometric mean concentration (GMC) > 0.1 IU/mL | At Week 4 after vaccination
  Vaccine cohort only
Proportion of participants with IgG serologic response to the tetanus toxoid with ≥ 4-fold increase in antibody GMC | At Week 4 after vaccination
  Vaccine cohort only
Pneumococcal opsonophagocytic assay (OPA) geometric mean titers (GMTs) | At Week 4 after vaccination
  Vaccine cohort only
Pneumococcal OPA geometric mean fold rise (GMFRs) | At Week 4 after vaccination
  Vaccine cohort only
Incidence of treatment-emergent adverse events (TEAEs) | At Week 4 after vaccination
  Vaccine cohort only
Incidence of serious adverse events (SAEs) | At Week 4 after vaccination
  Vaccine cohort only
Incidence of AEs leading to discontinuation | At Week 4 after vaccination
  Vaccine cohort only
Incidence of vaccine-specific AEs | At Week 4 after vaccination
  Vaccine cohort only

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (290):
- United States (101):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Local Institution - 0278, Birmingham, Alabama
  - Alliance Dermatology and Mohs Center - Phoenix, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Synexus - Orange Grove Family Practice, Tucson, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Northwest Arkansas Clinical Trials Center, PLLC, Rogers, Arkansas
  - Local Institution - 0046, Fountain Valley, California
  - Local Institution - 0206, Fresno, California
  - Local Institution - 0017, Irvine, California
  - Interspond - Long Beach Clinical Trials, Long Beach, California
  - Dermatology Research Associates - Los Angeles, Los Angeles, California
  - Local Institution - 0236, Los Angeles, California
  - University of California San Diego Health Systems, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - University Dermatology Group, San Diego, California
  - Local Institution - 0094, San Luis Obispo, California
  - Clinical Science Institute, Santa Monica, California
  - NorthBay Clinical Research, Santa Rosa, California
  - Synexus - Santa Rosa, Santa Rosa, California
  - Local Institution - 0042, Sherman Oaks, California
  - Care Access Research - Walnut Creek, Walnut Creek, California
  - New England Research Associates, Bridgeport, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Local Institution - 0170, Boca Raton, Florida
  - ERN - Accel Research Sites, DeLand, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - LCC Medical Research, Miami, Florida
  - International Dermatology Research, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Local Institution - 0216, Miami, Florida
  - Interspond - Savin Medical Group, Miami Lakes, Florida
  - Local Institution - 0007, Miami Lakes, Florida
  - Local Institution - 0198, Port Orange, Florida
  - Local Institution - 0233, Tampa, Florida
  - Local Institution - 0008, Tampa, Florida
  - Local Institution - 0013, Marietta, Georgia
  - Local Institution - 0235, Sandy Springs, Georgia
  - Treasure Valley Dermatology & Skin Cancer Center, Meridian, Idaho
  - Springfield Clinic, Springfield, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Clinical Research Advantage - Evansville - South Kenmore Drive, Evansville, Indiana
  - Dawes Fretzin Dermatology Group, Indianapolis, Indiana
  - Local Institution - 0020, Plainfield, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Local Institution - 0040, Louisville, Kentucky
  - Shondra L. Smith, M.D., Lake Charles, Louisiana
  - Clinical Trials of America - Monroe, Monroe, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Local Institution - 0291, Boston, Massachusetts
  - Ora, Chestnut Hill, Massachusetts
  - Local Institution - 0234, Methuen, Massachusetts
  - DermCare Experts, Quincy, Massachusetts
  - David Fivenson MD Dermatology, Ann Arbor, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Local Institution - 0025, Troy, Michigan
  - Associated Skin Care Specialists - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Washington University School of Medicine - West County Dermatology, St Louis, Missouri
  - Clinical Research Consortium - Las Vegas, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Local Institution - 0016, East Windsor, New Jersey
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Local Institution - 0058, New York, New York
  - Local Institution - 0218, Stony Brook, New York
  - Montefiore Medical Center - Bronx, The Bronx, New York
  - PMG Research of Cary, Cary, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Radiant Research - Columbus, Columbus, Ohio
  - ClinOhio Research Services, Columbus, Ohio
  - Local Institution - 0176, Fairborn, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Local Institution - 0167, Portland, Oregon
  - Local Institution - 0009, Portland, Oregon
  - Local Institution - 0045, Exton, Pennsylvania
  - Local Institution - 0282, Pittsburgh, Pennsylvania
  - Radiant Research - Anderson, Anderson, South Carolina
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Local Institution - 0037, Greer, South Carolina
  - Coastal Carolina Research Center - Mount Pleasant, North Charleston, South Carolina
  - Local Institution - 0004, Rapid City, South Dakota
  - Rivergate Dermatology - Main Office, Goodlettsville, Tennessee
  - Clinical Research Solutions - Jackson, Jackson, Tennessee
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - The Skin Wellness Center, Knoxville, Tennessee
  - Local Institution - 0006, Arlington, Texas
  - Bellaire Dermatology, Bellaire, Texas
  - Local Institution - 0015, Dallas, Texas
  - Local Institution - 0195, Dallas, Texas
  - Local Institution - 0030, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies - Texas Medical Center, Houston, Texas
  - Austin Institute for Clinical Research - Pflugerville, Pflugerville, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Interspond - Acclaim Dermatology, Sugar Land, Texas
  - Interspond - Houston Center for Clinical Research, Sugar Land, Texas
  - Center for Clinical Studies - Webster, Webster, Texas
  - Local Institution - 0265, Seattle, Washington
- Australia (12):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Local Institution - 0246, Darlinghurst, New South Wales
  - St. George Dermatology & Skin Care Centre, Kogarah, New South Wales
  - Local Institution - 0250, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Local Institution - 0241, Woolloongabba, Queensland
  - North Eastern Health Specialists, Hectorville, South Australia
  - Local Institution - 0245, Box Hill, Victoria
  - Skin and Cancer Foundation, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Local Institution - 0251, Parkville, Victoria
  - Local Institution - 0247, Perth, Western Australia
- Canada (22):
  - Beacon Dermatology, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - SkinFit MD Laser and Cosmetic Clinic, Surrey, British Columbia
  - Local Institution - 0152, Vancouver, British Columbia
  - Wiseman Dermatology Research, Winnipeg, Manitoba
  - CCA Medical Research, Ajax, Ontario
  - Mediprobe Research, London, Ontario
  - Local Institution - 0090, London, Ontario
  - Lynderm Research, Markham, Ontario
  - DermEdge, Mississauga, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Office of Dr. Niakosari Firouzeh, North York, Ontario
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario
  - Local Institution - 0088, Peterborough, Ontario
  - Local Institution - 0082, Richmond Hill, Ontario
  - Toronto Dermatology Centre, Toronto, Ontario
  - Local Institution - 0132, Toronto, Ontario
  - Kim Papp Clinical Research, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Docteur David Gratton Dermatologue, Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
  - Local Institution - 0258, Québec, Quebec
- China (10):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Wuhan, Hubei
  - Local Institution - 0312, Nanjing, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Dalian, Liaoning
  - Local Institution, Taiyuan, Shan1xi
  - Local Institution - 0292, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Hangzhou, Zhejiang
- Czechia (7):
  - Nemocnice Jihlava, Jihlava
  - Nemocnice Novy Jicin a.s., Nový Jičín
  - Local Institution - 0163, Olomouc
  - Local Institution - 0165, Ostrava
  - Clintrial, Prague
  - Sanatorium profesora Arenbergera, Prague
  - Krajska zdravotni - Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- Local Institution - 0279, Tampere, Finland
- Centre Hospitalier Universitaire de Nice Hopital lArchet, Nice, France
- Germany (9):
  - Licca Clinical Research Institute, Augsburg
  - Hautarztpraxis Dr. Niesmann & Dr. Othlinghaus, Bochum
  - Hautarztpraxis Dr. Beatrice Gerlach, Dresden
  - Synexus Frankfurt Clinical Research, Frankfurt am Main
  - Local Institution - 0263, Hamburg
  - Dermakiel - Allergie Und Haut Centrum, Kiel
  - Praxis Dr. Beate Schwarz, Langenau
  - Praxis Dr. med. Wilfried Steinborn, Straubing
  - CentroDerm Privatklinik, Wuppertal
- Hungary (10):
  - Qualiclinic Egeszsegugyi Szolgaltato es Kutatasszervezo Kft., Budapest
  - Synexus Magyarorszag, Budapest
  - Semmelweis Egyetem, Budapest
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato - Debrecen Affiliated Site, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato - Gyula, Gyula
  - Josa Andras Oktatokorhaza - Szabolcs Szatmar-Bereg Megyei Onkormanyzat, Nyíregyháza
  - Local Institution - 0151, Pécs
  - Allergo-Derm Bakos, Szolnok
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato - Zalaegerszeg, Zalaegerszeg
- Israel (3):
  - Local Institution - 0237, Haifa
  - Local Institution, Petah Tikva
  - Local Institution, Ramat Gan
- Japan (24):
  - Local Institution - 0065, Nagoya, Aichi-ken
  - Local Institution - 0069, Fukuoka, Fukuoka
  - Sapporo Skin Clinic, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Tokai University Hospital, Isehara, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Local Institution - 0075, Yokohama, Kanagawa
  - Local Institution - 0076, Nankoku, Kochi
  - Local Institution - 0066, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Local Institution - 0072, Matsumoto, Nagano
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Local Institution - 0061, Itabashi-Ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Local Institution - 0062, Shinagawa, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Japan Community Health Care Organization Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Local Institution - 0096, Kumamoto
  - Local Institution - 0093, Kyoto
  - Local Institution - 0073, Osaka
  - Local Institution - 0067, Osaka
- New Zealand (2):
  - Local Institution, Mount Cook
  - Local Institution, Tauranga
- Poland (32):
  - Local Institution - 0138, Warsaw, Masovian Voivodeship
  - Local Institution - 0104, Bialystok
  - ZDROWIE OSTEO-MEDIC s.c. Lidia i Artur Racewicz, Agnieszka i Jerzy Supronik, Bialystok
  - ClinicMed Daniluk Nowak Spolka Jawna, Bialystok
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag
  - Local Institution - 0149, Gdansk
  - Synexus Polska Oddzial w Gdyni, Gdynia
  - Zespol Naukowo-Leczniczy Iwolang, Iwonicz-Zdrój
  - Synexus - Katowice, Katowice
  - Krakowskie Centrum Medyczne, Krakow
  - Pratia MCM Krakow, Krak
  - Centrum Terapii Wspolczesnej, Lodz
  - Local Institution - 0114, Lodz
  - Local Institution - 0144, Lodz
  - Centrum Medyczne All-Med, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej MED-LASER, Lublin
  - Miejski Szpital Zespolony w Olsztynie, Olsztyn
  - DermoDent - Centrum Medyczne Czajkowscy, Osielsko
  - Local Institution - 0103, Poznan
  - Solumed Centrum Medyczne, Poznan
  - ETG - Siedlce, Siedlce
  - Local Institution - 0113, Skierniewice
  - Local Institution - 0125, Torun
  - Clinical Research Group, Warsaw
  - High-Med Przychodnia Specjalistyczna, Warsaw
  - Local Institution - 0119, Warsaw
  - Local Institution - 0324, Warsaw
  - Local Institution - 0111, Warsaw
  - Local Institution - 0137, Wroc?aw
  - dermMedica Sp. z o.o., Wroclaw
  - Local Institution - 0124, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Local Institution - 0289, San Juan, Puerto Rico
- Russia (13):
  - Local Institution - 0172, Kazan'
  - Local Institution - 0187, Krasnodar
  - Local Institution - 0171, Moscow
  - Local Institution - 0175, Moscow
  - Local Institution - 0169, Moscow
  - Local Institution - 0190, Ryazan
  - Local Institution - 0179, Saint Petersburg
  - Local Institution - 0182, Saint Petersburg
  - Local Institution - 0201, Saint Petersburg
  - Local Institution - 0202, Saratov
  - Local Institution - 0184, Smolensk
  - Local Institution - 0222, Yaroslavl
  - Local Institution - 0178, Yekaterinburg
- South Korea (13):
  - Local Institution - 0306, Seongnam-si, Gyeonggi-do
  - Local Institution, Bucheon-si
  - Local Institution - 0054, Busan
  - Local Institution, Goyang-si
  - Local Institution - 0310, Gwangju
  - Local Institution, Hwaseong-si
  - Local Institution, Incheon
  - Local Institution - 0051, Seongnam-si
  - Local Institution, Seoul
  - Local Institution - 0305, Seoul
  - Local Institution - 0055, Seoul
  - Local Institution - 0053, Seoul
  - Local Institution, Suwon
- Spain (9):
  - Local Institution - 0223, Alcorcón
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Local Institution - 0230, Barakaldo
  - Local Institution - 0225, Córdoba
  - Local Institution - 0226, Las Palmas de Gran Canaria
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital de Manises, Manises
  - Local Institution - 0227, Málaga
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
- Sweden (3):
  - Ladulaas Kliniska Studier, Borås
  - ProbarE i Lund, Lund
  - Local Institution - 0186, Solna
- Taiwan (4):
  - Local Institution - 0079, Kaohsiung City
  - Local Institution - 0297, Kaohsiung City
  - Local Institution, Taipei
  - Local Institution - 0153, Taipei
- United Kingdom (13):
  - MAC Clinical Research - Cannock, Cannock
  - Synexus - Lancashire Clinical Research Centre, Chorley
  - Synexus - Manchester Clinical Research Centre, Chorley
  - Synexus - Merseyside Clinical Research Centre, Chorley
  - Mounts Bay Medical, Cornwall
  - The Dudley Group NHS Foundation Trust, Dudley
  - Local Institution - 0212, Durham
  - MAC Clinical Research - Blackpool, Lancashire
  - Burbage Surgery, Leicestershire
  - Guys and Saint Thomas NHS Foundation Trust, London
  - MAC Clinical Research - Manchester, Manchester
  - Salford Royal NHS Foundation Trust, Manchester
  - Local Institution - 0209, Prescot

REFERENCES:
- [Derived] Armstrong AW, Kircik L, Stein Gold L, Strober B, De Oliveira CHMC, Vaile J, Jou YM, Daamen C, Scharnitz T, Lebwohl M. Deucravacitinib: Laboratory Parameters Across Phase 3 Plaque Psoriasis Trials. Dermatol Ther (Heidelb). 2025 Apr;15(4):1025-1035. doi: 10.1007/s13555-025-01362-w. Epub 2025 Mar 20. PMID 40113724
- [Derived] Morita A, Imafuku S, Tada Y, Okubo Y, Habiro K, Tsuritani K, Banerjee S, Hoyt K, Kisa RM, Ohtsuki M. Deucravacitinib in plaque psoriasis: Safety and efficacy through 3 years in Japanese patients in the phase 3 POETYK PSO-1, PSO-4, and LTE trials. J Dermatol. 2025 May;52(5):761-772. doi: 10.1111/1346-8138.17685. Epub 2025 Mar 11. PMID 40066907
- [Derived] Armstrong AW, Lebwohl M, Warren RB, Sofen H, Imafuku S, Ohtsuki M, Spelman L, Passeron T, Papp KA, Kisa RM, Vaile J, Berger V, Vritzali E, Hoyt K, Colombo MJ, Scotto J, Banerjee S, Strober B, Thaci D, Blauvelt A. Safety and Efficacy of Deucravacitinib in Moderate to Severe Plaque Psoriasis for Up to 3 Years: An Open-Label Extension of Randomized Clinical Trials. JAMA Dermatol. 2025 Jan 1;161(1):56-66. doi: 10.1001/jamadermatol.2024.4688. PMID 39602111
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04036435.html